CLINICAL TRIAL: NCT06302712
Title: Cultural Adaptation and Evaluation of Traditional Islamically Integrated Psychotherapy for Muslim With OCD in Pakistan: A Mixed-Method Study.
Brief Title: Traditional Islamically Integrated Psychotherapy for Muslims With OCD in Pakistan
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: International Islamic University Malaysia (Other)
Collaborators: Foundation University Islamabad (Other)
Responsible Party: Principal Investigator, Jamilah Hanum Abdul Khaiyom, PhD, Assistant Professor., International Islamic University Malaysia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TIIP
Record Dates: First submitted 2024-03-04; First posted 2024-03-12 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Obsessive-Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental)
  Interventions: Behavioral: Traditional Islamically Integrated Psychotherapy
- TAU (No Intervention)

INTERVENTIONS:
Behavioral: Traditional Islamically Integrated Psychotherapy — Traditional Islamically Integrated Psychotherapy for OCD. We will be using the culturally adapted module of TIIP that is translated into the Urdu language for Pakistan Muslims with OCD. The treatment module is mainly based on four domains Nafs (Behavior), Ihsas (Emotions), Aql (Thought), and Ruh (Spirituality). The session will be conducted in an individual format, with eight sessions, and the intervention will be conducted by a certified therapist in TIIP.
  Arms: Intervention

SUMMARY:
The current study aims to determine the effectiveness of the first culturally adapted Traditional Islamically Integrated Psychotherapy (TIIP) for Muslims with OCD in Pakistan along with the module effectiveness in reducing OCD symptoms with comorbidities like anxiety, depression, stress, thought control, thought-action fusion, and enhancing the spiritual quality of life of participants.

ELIGIBILITY:
Inclusion Criteria:

* The client diagnosed with OCD according to DSM-5-TR.
* The minimum score on Y-BOCS is 08 (i.e., indicating moderate level of symptoms)
* The age range is from 18 to 40 years
* The client has a minimum of eight years of formal education

Exclusion Criteria:

* The client is having a comorbid diagnosis of severe psychiatric illness (e.g., psychotic disorders, personality disorder, substance use disorder, neurocognitive disorder)
* The client is having a comorbidity of chronic physical illness
* The client refused to sign the informed consent form,
* The client has experience undergoing manualized faith-based CBT

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-11-30 (Estimated)

PRIMARY OUTCOMES:
Yale Brown Obsessive Compulsive Scale | 8 weeks
  Yale Brown Obsessive Compulsive is a 10-item self-report scale developed to assess the severity of both obsession and compulsion.
  Minimum score is 0 and maximum score is 40. The higher the scores mean the worst outcome.
  Cut-off Scores:
  0-7 (sub-clinical) 8-15 (Mild) 16-23 (Moderate) 24-31 (severe) 32-40 (Extrerme)

SECONDARY OUTCOMES:
Depression, Stress, Anxiety | 8 Weeks.
  Depression, Stress, Anxiety is measured through scale
  Minimum score is 0 and maximum score is 42. The higher the scores mean the worst outcome.
  Cut-off scores for each subscales.
  Stress:
  0-10 (normal) 11-18 (mild) 19-26 (moderate) 27-34 (severe) 35-42 (Extremely severe)
  Anxiety:
  0-6 (normal) 7-9 (mild) 10-14 (moderate) 15-19 (severe) 20-42 (Extremely severe)
  Depression:
  0-9 (normal) 10-12 (mild) 13-20 (moderate) 21-27 (severe) 28-42 (Extremely Severe)
Thought Action Fusion | 8 weeks
  Thought Action Fusion is measured with the help of Thought Action Fusion Scale
  Minimum score is 0 and maximum score is 76. The higher the scores mean the worst outcome.
Thought Control | 8 weeks
  Thought Control is measured with the help of Thought Control Questionnaire
  Minimum score is 30 and maximum score is 120. The higher the scores mean the worst outcome.
Spiritual Quality | 8 weeks
  Spiritual Quality is measured with the help of World Health Organization Quality of Life Spirituality, Religiousness and Personal Beliefs Scale
  Minimum score is 9 and maximum score is 45. The higher the scores mean the worst outcome.